CLINICAL TRIAL: NCT07181421
Title: Impact of Tissue Flossing and Therapeutic Exercises in Patient With Knee Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/05
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Knee Osteoarthristis
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tissue Flossing and Therapeutic Exercises (Experimental): Detailed of tissue flossing and therapeutic exercises.: The floss band will be kept on for 2 minutes, and during this time, the patient will perform the exercises with progression. After each 2-minute flossing session, the patient will rest for 2 minutes.
  Interventions: Procedure: Tissue flossing with Therapeutic exercises
- Therapeutic Exercises only (Active Comparator): Isometric Knee Extension - Standing Hamstring Curl - Wall Squats - Leg Press Against Wall
  Interventions: Procedure: Therapeutic Exercises

INTERVENTIONS:
Procedure: Tissue flossing with Therapeutic exercises — Isometric Knee Extension - Standing Hamstring Curl - Wall Squats - Leg Press Against Wall. The Red TheraBand from Thera Tool (2m * 5cm * 1.3mm) will be used. The band will be wrapped starting from the tibial tuberosity and extending to 5 cm above the femoral epicondyle. Care will be taken to ensure that the patella remains uncovered.
  * The band will be wrapped with 50% tension and 50% overlap.
  * Flossing Duration: The floss band will be kept on for 2 minutes, and during this time, the patient will perform the exercises mentioned above. The number of repetitions for each exercise will depend on the patient's tolerance level, with a reference of 10 repetitions per exercise (based on similar tissue flossing protocols, though adapted for knee OA patients).
  Arms: Tissue Flossing and Therapeutic Exercises
Procedure: Therapeutic Exercises — Isometric Knee Extension - Standing Hamstring Curl - Wall Squats - Leg Press Against Wall.
  Arms: Therapeutic Exercises only

SUMMARY:
Knee osteoarthritis (OA) is a common degenerative joint disease that primarily affects individuals aged 40 years and older, and results in painful symptoms along with limited range of motion (ROM) and muscle weakness(1). Therapeutic exercise covers a range of targeted physical activities that directly aim to improve muscle strength, neuromotor control, joint range of motion and aerobic fitness. One of the main aims of exercise is to improve muscle strength, given that weakness is common in knee OA. Exercise, especially isometric ROM exercises and step-ups as therapeutic exercise, are very important in OA patients, because they not only maintain the activity of the joint but also treat the pain and strengthen the joint (2).Use of tissue flossing, in which an elastic band is wrapped around muscles and joints to enhance blood flow and reduce pain(3).It has been on the rise as an adjunct to rehabilitation, but its efficacy when combined with therapeutic exercise is not well-known. The objective of this non-blinded randomized controlled trial is to compare the effects of tissue flossing combined with therapeutic exercises versus therapeutic exercises alone on pain, ROM, and muscle strength in patients with knee OA. The study will be conducted over a period of 4 weeks, with two sessions per week at Sheikh Khalifa Bin Zayed Hospital, Quetta. Initially, participants aged 40-70 years with diagnosed Grade 1,2and 3 knee OA will be screened for eligibility based on inclusion and exclusion criteria. Eligible participants will be informed about the study objectives and procedures, and written informed consent will be obtained. Participants will then be randomly allocated into two groups using the envelope method for group randomization. Baseline assessment will include knee ROM measurement, muscle strength assessment using Manual Muscle Testing (MMT), pain evaluation using the Numeric Pain Rating Scale (NPRS), Group A will receive tissue flossing in addition to therapeutic exercises, while Group B will receive only therapeutic exercises. All outcome measures will be reassessed after 4 weeks of intervention to evaluate the effects of the intervention. Data will be entered and analyzed using SPSS v.22.

DETAILED DESCRIPTION:
Knee Osteoarthritis (OA) is a chronic degenerative joint disorder characterized by the breakdown of articular cartilage, synovial inflammation, and structural changes in subchondral bone, leading to pain, stiffness, and functional limitations (1). Knee OA, the most prevalent form of OA, significantly affects mobility and quality of life, especially in individuals with sedentary lifestyles or obesity. According to the Global Burden of Disease (GBD) report, knee OA accounts for a substantial proportion of disability-adjusted life years (DALYs), with high body mass index (BMI) identified as a major risk factor. By 2050, an estimated 642 million individuals are expected to suffer from knee OA, highlighting the urgent need for effective therapeutic interventions(4).Non pharmacological approaches, particularly therapeutic exercises, remain central to knee OA management.

Even a few degrees of extension or flexion loss can affect function and cause pain. The opposite, normal knee must be examined to establish a baseline for normal ROM. In patients with knee OA, most nonoperative rehabilitation programs concentrate on increasing strength, which is difficult to achieve when any ROM loss is present. The Shelbourne Knee Center ROM-based rehabilitation program emphasizes normalizing knee extension, followed by improving flexion and then strength. This ROM-based rehabilitation program has been effective for improving ROM, pain, symptoms, and function in patients with OA, and 76% were prevented from undergoing TKA surgery(5).

Exercise, particularly isometric range of motion (ROM) exercises and step-ups, plays a crucial role in managing osteoarthritis (OA). These exercises help maintain joint activity, alleviate pain, and strengthen the joint. For instance, a study published in Cures demonstrated that isometric strengthening exercises significantly reduced pain intensity and improved functional ability in patients with knee osteoarthritis(6). The meta-analysis finding indicates that isometric exercise is an effective physical therapy for treating KOA. It significantly reduces pain, improves physical function, and enhances muscle strength in KOA patients making it a valuable therapeutic option(7). Progressive resistance training, where the resistance is progressively increased to maintain relative intensity, can lead to significant improvements in older adults with knee OA by ameliorating sarcopenic changes and by improving the strength and function of the surrounding connective tissue, which is often damaged by the disease.(21)(22) However, despite their proven benefits, a significant proportion of patients continue to experience pain and functional limitations, necessitating the exploration of complementary interventions to optimize outcomes. Tissue flossing, a technique introduced by Dr. Kelly Starrett in 2014, has emerged as a novel adjunct therapy. Tissue flossing was first proposed by Starrett and Cordoza (2015), who suggested that flossing can increase the range of motion and/or performance (strength ), speed up recovery, and decrease pain caused by various disease or injuries. This intervention involves the application of elastic bands with controlled compression around the joint or muscle, followed by functional movements. Konrad., et al. in 2021 states that the mechanism of tissue flossing is hypothesized to enhance blood flow, reduce fascial adhesions, promote lymphatic drainage, and improve joint mobility (8). Pavlu D., et al. in 2021 indicate that tissue flossing is effective in reducing pain, improving range of motion (ROM), and enhancing functional capacity (9). A study by Driller.,et al. in 2017 states Flossing involves the mechanism of the ischemic preconditioning afterwards the reperfusion of the blood into the flossed area could be associated with subsequent increases in growth hormone, catecholamine responses, increased muscle force and contractility and increased efficiency of excitation-contraction coupling in the muscles (10). The mechanisms behind tissue flossing can also be described as facial shearing where the compression together with movement alter the relationship with the fascia and the neuromuscular system(8). The choice of Kallgren-Lawrence Grades 1,2 and 3 for my study is supported by literature that indicates their physical therapy suitability. Tuna et al. (2022) reported that physical therapy with exercises benefited pain relief at all grades of peripheral knee osteoarthritis (OA).In addition, the majority of radiological OA patients are likely to have KL Grade II and III ranging from 12% to 17% (12). This grade is at a moderate disease severity level, which is great for studying the impacts of tissue flossing. These early stages of the disease are more common and easier to treat, therefore it is beneficial to prioritize these grades to maximize function. A systematic review showed that the effects of floss band could lead to noticeable improvement in the general population and patients. (8). This study aims to evaluate the combined effects of tissue flossing and therapeutic exercises on pain relief, ROM, and muscle strength in patients with knee OA. By addressing gaps in the current literature, the findings of this study may provide innovative and clinically relevant strategies for managing knee OA, thereby improving patient outcomes and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40-70 years with diagnosed knee OA (Grades 1 and 2). Unilateral knee OA or if bilateral OA is present, only the more symptomatic knee (Grade 1 or 2) Willingness to comply with the intervention protocol. Both Genders

Exclusion Criteria:

* Higher grade 3 and 4 knee OA. Recent knee surgeries Soft tissue injury of lower limb less than six months prior to the study Neurological or cardiovascular conditions contraindicating exercise Ongoing participation in another knee Rehabilitation program Latex allergy or Skin diseases varicose veins and Thrombosis Diabetic Neuropathy Fractures and open wounds.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Knee Pain | 4 weeks
  Numeric pain rating scale will be used to measure knee pain
Knee Range of Motion | 4 weeks
  Goniometer willl be used to measure knee range of motion
Knee Muscle Strength | 4 weeks
  Manual Muscle Testing will be used for knee muscle strength

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University Islamabad, Islamabad, Punjab Province, Pakistan